CLINICAL TRIAL: NCT02651272
Title: The Safety and Efficacy of Macitentan for Treatment of Pulmonary Hypertension in Sickle Cell Disease
Brief Title: Macitentan in Pulmonary Hypertension of Sickle Cell Disease
Acronym: MENSCH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll IRB approved sample of participants.
Sponsor: Boston University (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-33165
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Hypertension; Sickle Cell Disease
Keywords: Pulmonary Hypertension; Sickle Cell Disease; Pulmonary Arterial Hypertension; Macitentan
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell; Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Masking Description: Study is Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- macitentan (Experimental): 10mg macitentan tablets, taken once daily (QD), by mouth (PO), for the treatment period lasting 16 weeks.
  Interventions: Drug: macitentan

INTERVENTIONS:
Drug: macitentan — 10mg macitentan tablets
  Other Names: opsumit

SUMMARY:
This is a pilot study to assess the safety and efficacy of macitentan in patients with pulmonary hypertension of sickle cell disease. This study will enroll approximately 10 subjects. Study participation for each subject will last approximately 24 weeks from screening to end of treatment follow-up.

DETAILED DESCRIPTION:
Background and Rationale:

Sickle cell disease (SCD) affects 250,000 births per year worldwide, with 70-80,000 patients currently residing in the US. Although classically thought of as a genetic hemoglobinopathy, most of the clinical complications are vascular in etiology and pulmonary manifestations are the primary cause of morbidity and mortality. Pulmonary hypertension (PH), one such pulmonary complication, occurs in 6-10.5% of SCD adults and is associated with a 60% four-year survival. No specific therapy for PH in SCD exists representing an area of intense clinical need in this field.

Clinical trials of pulmonary vasodilator medications in PH of SCD have been problematic. There have been no randomized placebo controlled trials of any traditional pulmonary arterial hypertension (PAH) medication completed in this population to date. Three randomized placebo-controlled trials have been undertaken previously. Two compared treatment with bosentan to placebo in SCD patients with right heart catheterization (RHC) -defined elevated pulmonary vascular resistance (PVR) with a normal pulmonary capillary wedge pressure (PCWP) (the ASSET-1 trial) or pulmonary venous hypertension (PVH) with a PVR > 100 dynes.sec/cm5 (the ASSET-2 trial). After the randomization of only 14 subjects in ASSET-1 and 12 patients in ASSET-2, the trials were prematurely terminated due to slow patient enrollment. Although very few patients were enrolled, there were no apparent toxicity issues. The third trial, Walk-PHaSST (Pulmonary Hypertension and Sickle Cell Disease with Sildenafil Therapy), compared the safety and efficacy of sildenafil to placebo in SCD patients with a TRV ≥2.7m/s. After 74 (of a targeted 132) subjects were enrolled, the study was prematurely discontinued due to an increase in serious adverse events in the sildenafil group, primarily hospitalization for pain.

There are a number of possible explanations for these failed trials:

1. The hemodynamics of PH in SCD reflect a spectrum of abnormalities. Approximately 40-50% of PH in SCD patients have hemodynamics similar to other forms of PAH; a mean pulmonary arterial pressure >25 mmHg, normal left-sided filling pressures (PCWP or left ventricular end diastolic pressure <15 mmHg) and an elevated PVR. But at least 50% of PH in SCD patients have at least some degree of PVH usually due to diastolic dysfunction of the left ventricle. How an elevated PVR is defined in PH of SCD is controversial. While typically in other forms of PAH, it is defined as 3 Wood units or 240 dynes.sec/cm5, this is reflective of a normal PVR of 120-160 dynes.sec/cm5. In SCD, the anemia-induced elevations in cardiac output observed in these patients produce a baseline PVR of 60-100 dynes.sec/cm5 suggesting that a PVR of 160 dynes.sec/cm5 or 2 Wood units may be a more appropriate value.
2. SCD is considered to be a rare disease in the US according to the NIH. As PAH of SCD probably only occurs in 2-4% of HbSS adults, many centers in the US will only have a few (<10) eligible patients for enrollment even under the best circumstances. SCD patients often have co-morbidities limiting their participation in clinical trials, which often decreases this number even further.
3. The epidemiology of PH in SCD has been evolving over the past 10-15 years. Numerous studies demonstrated an elevated pulmonary artery systolic pressure (PASP) by echocardiography reflected by an elevated tricuspid regurgitant jet velocity (TRV) was present in 1/3 of HbSS and 10-28% of HbSC adults. However, an elevated TRV only has approximately a 25% positive predictive value for PH in SCD. The need for a right heart catheterization to confirm a diagnosis of PH in SCD has only been gaining clinical acceptance over the past few years and when the prior clinical trials were conducted, this was not a standard part of the PH workup in these patients.

Given the serious limitations of the randomized trials, our clinical guidelines committee decided that its judgments regarding whether targeted PAH therapy is indicated in SCD patients with an elevated PVR and normal PCWP should be informed by indirect evidence from Group 1 PAH populations and our own clinical experience. In Group 1 PAH patients, it has been well-established by meta-analyses of randomized trials that targeted PAH therapy consistently improves exercise capacity, functional status, symptoms, cardiopulmonary hemodynamics and outcome. This indirect evidence is supported by four case series in which SCD patients with RHC-confirmed pre-capillary PH received targeted PAH therapy with bosentan, sildenafil, and/or epoprostenol. Targeted PAH therapy was associated with improvement in exercise capacity, with the six minute walk distance increasing 41 to 144 m beyond baseline. There were also improvements in the mean pulmonary artery pressure (PAP), PVR, and cardiac index, although these parameters were measured in only a few patients. The magnitude of the benefits was greatest among symptomatic patients. The most common adverse effects were headache (15%) and peripheral edema (21%); transaminase elevation was reported in 14% of patients during endothelin receptor antagonist therapy. Based upon these results and the increased morbidity associated with sildenafil use, we are weakly recommending a trial of either a prostanoid or an endothelin receptor antagonist for select patients with SCD who have a RHC-confirmed marked elevation of their PVR, normal PCWP, and related symptoms.

The FDA approval of macitentan for treatment of PAH represents a unique opportunity for study of the use of this medication in SCD. Endothelin-1 has long been established as an important mediator of vasoconstriction in SCD [19, 20] and more recent studies have implicated a role for this molecule in mouse models of PH in SCD [21]. PH and an elevated TRV are both independent risk factors for mortality in SCD [1, 2, 9, 22] and, as the median age of death of SCD patients is in the 5th decade irrespective of a PH diagnosis, the possibility of therapeutically altering this outcome is of key importance in this disease. With the publication of the American Thoracic Society sponsored clinical guidelines for the diagnosis and treatment of PH in SCD (additionally endorsed by the Pulmonary Hypertension Association and the American College of Chest Physicians), the timing for re-addressing the possibility of a clinical trial of a PAH therapy in this population perfect. We propose to utilize the information gathered from the trials which proceeded it to specifically design a clinical trial using macitentan to treat the SCD patients most likely to respond to this therapy; those with PAH-like hemodynamics without co-existent left-sided heart disease.

Hypotheses:

1. Macitentan will be safe for treatment in patients with PAH of sickle cell disease
2. Macitentan will improve hemodynamics, exercise capacity and quality of life in patients with pre-capillary pulmonary hypertension of sickle cell disease
3. Long-term use of macitentan will improve survival in patients with sickle cell disease and pulmonary hypertension

Study Design:

To conduct a 16 week prospective open-label Phase II clinical trial of macitentan in SCD patients with hemodynamics consistent with pulmonary arterial hypertension.

We plan to enroll 10 patients in this study. All enrolled patients will be treated with 10 mg macitentan daily for the entire treatment period.

The study is comprised of the three consecutive periods:

Screening Period/Baseline Studies:

This period will be up to 30 days in duration, commencing with the first screening visit and completing with the start of study medication.

Treatment Period:

This will begin at Visit 2, the baseline visit and will continue until the end of 16 weeks of therapy or earlier in the case of premature stoppage of treatment. During this period, there will be a safety assessment at the first visit followed by visits to assess safety and efficacy at weeks 4, 8, 12 and 16.

Post-Treatment Study Period:

This will last 30 days after the completion of the treatment period and will allow for additional assessment of medication safety.

Screening Period:

After obtaining informed consent, the patient will undergo the screening protocol which includes assessment of baseline demographics (sex, age, race, ethnicity, height, and body weight), as well as an assessment of why the female patients are not of child-bearing potential as appropriate. The following data will be obtained:

1. Medical history- To include:

   1. SCD related complications (stroke, AVN, priapism, lower extremity ulcers etc.)
   2. Frequency of vaso occlusive crises and hospitalizations
   3. Frequency of blood transfusions
   4. History and frequency of acute chest syndrome
   5. History of thromboembolic disease
   6. History of congestive heart failure
   7. History of asthma
   8. History of systemic hypertension
   9. History of proteinuria
   10. History of chronic kidney disease
   11. Echocardiogram and any data from previous echos over past 12 months
   12. Pulmonary function data from the prior 12 months
2. Concomitant Medication Use - All medications will be recorded. Hydroxyurea use will be assessed in all subjects.
3. Physical Examination and Vital Signs
4. 12 lead electrocardiogram
5. Laboratory Testing: Complete blood counts, blood chemistries including BUN and creatinine, liver function testing, markers of hemolysis (lactate dehydrogenase, total and indirect bilirubin, AST, reticulocyte counts), urinalysis, urine pregnancy test and NT-pro-BNP levels.
6. WHO Functional Class
7. 6 minute walk test and Borg Dyspnea Score
8. Short form (SF)-36 questionnaire
9. Right Heart Catheterization (can be done up to 12 weeks prior to initiation of study medication).

Baseline Visit (Day 1):

1. Medical History
2. Concomitant Medication Usage
3. Physical Examination and Vital Signs
4. Laboratory and Pregnancy Testing
5. WHO functional class
6. 6 minute walk test and Borg Dyspnea Score
7. SF-36 questionnaire

Week 4 visit:

1. Physical Examination and Vital Signs
2. Laboratory and Pregnancy Testing
3. Assessment of Adverse Events

Week 8 Visit:

1. Medical History
2. Concomitant Medication Usage
3. Physical Examination and Vital Signs
4. Laboratory and Pregnancy Testing
5. WHO functional class
6. 6 minute walk test and Borg Dyspnea Score
7. SF-36 questionnaire
8. Assessment of Adverse Events

Week 12:

1. Physical Examination and Vital Signs
2. Laboratory and Pregnancy Testing
3. Assessment of Adverse Events

Week 16:

1. Medical History
2. Concomitant Medication Usage
3. Physical Examination and Vital Signs
4. Laboratory and Pregnancy Testing
5. WHO functional class
6. 6 minute walk test and Borg Dyspnea Score
7. SF-36 questionnaire
8. Assessment of Adverse Events
9. 12 lead electrocardiogram
10. Right heart catheterization
11. Echocardiogram

Post-Treatment Follow-Up Visit:

1) Assessment of Adverse Events

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of sickle cell disease (HbSS, HbSC, HbS- β+ or 0) confirmed by hemoglobin electrophoresis
2. Provision of informed consent
3. Suspicion of Pulmonary Hypertension by echocardiography within the last 6 months (RVSP > 40mmHg or a TRV > 3.0 m/sec) or diagnosis of Pulmonary Hypertension by cardiac catheterization within the last 12 months (mean Pulmonary Artery Pressure [PAP] ≥25 mmHg at rest). Left ventricular ejection fraction > 50%.
4. Right heart catheterization which demonstrates the following:

   1. mean pulmonary arterial pressure [mPAP] > 25 mmHg
   2. pulmonary artery occluded pressure [PAOP] or LVEDP < 15 mmHg
   3. PVR > 160 dynes-sec/cm5 or 2 Wood Units
5. Age > 18 years
6. NYHA Class II or III by symptoms
7. Six minute walk distance (6MWD) > 150 meters and < 450 meters
8. A woman of child-bearing potential is eligible only if the following applies:

   1. Negative pre-treatment serum pregnancy test and agreement to monthly tests
   2. Use of two highly effective methods of contraception if not truly abstinent with a male partner OR permanent female sterilization has been performed.
9. May be on background therapy or may be treatment naïve.

Exclusion Criteria:

1. Current pregnancy or lactation
2. Any one of the following medical conditions:

   1. Stroke within the last 6 weeks
   2. New diagnosis of pulmonary embolism within the last 3 months
   3. Clinically significant laboratory abnormalities, including, but not limited to: Positive Hepatitis B surface antigen or Hepatitis C antibody, Positive HIV test, Serum alanine aminotransferase (ALT) greater than or equal to 2.0 x ULN, Serum creatinine greater than or equal to 2.5mg/dL (or calculated creatinine clearance less than or equal to 30mL/min).
   4. Hospitalization within the prior 4 weeks for a vasoocclusive crisis or acute chest syndrome
   5. Any unstable (acute or chronic) condition that in the opinion of the investigator will prevent completion of the study
3. Evidence of diastolic dysfunction of the left ventricle as defined by a mPAP > 25 mmHg and PCWP or LVEDP > 15 mmHg by right heart catheterization with a normal left ventricular ejection fraction by echocardiogram or MUGA.
4. Left ventricular ejection fraction < 50% of significant ischemic, valvular or constrictive heart disease
5. Acute or chronic impairment (other than dyspnea) limiting the ability to comply with study requirements (particularly the 6MWT) e.g. symptomatic hip osteonecrosis
6. Active therapy with an IV prostacyclin
7. Subjects who are taking other investigational medications at the time of the study
8. Clinically significant psychiatric, addictive (defined by DSM-IV criteria), neurologic disease or condition that, in the opinion of the Investigator, would compromise his/her ability to give informed consent, participate fully in this study, or prevent adherence to the requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07; Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Klings, MD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share IPD.

REFERENCES:
- [Background] Mehari A, Gladwin MT, Tian X, Machado RF, Kato GJ. Mortality in adults with sickle cell disease and pulmonary hypertension. JAMA. 2012 Mar 28;307(12):1254-6. doi: 10.1001/jama.2012.358. No abstract available. PMID 22453563
- [Background] Parent F, Bachir D, Inamo J, Lionnet F, Driss F, Loko G, Habibi A, Bennani S, Savale L, Adnot S, Maitre B, Yaici A, Hajji L, O'Callaghan DS, Clerson P, Girot R, Galacteros F, Simonneau G. A hemodynamic study of pulmonary hypertension in sickle cell disease. N Engl J Med. 2011 Jul 7;365(1):44-53. doi: 10.1056/NEJMoa1005565. PMID 21732836
- [Background] Fonseca GH, Souza R, Salemi VM, Jardim CV, Gualandro SF. Pulmonary hypertension diagnosed by right heart catheterisation in sickle cell disease. Eur Respir J. 2012 Jan;39(1):112-8. doi: 10.1183/09031936.00134410. Epub 2011 Jul 20. PMID 21778170
- [Background] Klings ES, Machado RF, Barst RJ, Morris CR, Mubarak KK, Gordeuk VR, Kato GJ, Ataga KI, Gibbs JS, Castro O, Rosenzweig EB, Sood N, Hsu L, Wilson KC, Telen MJ, Decastro LM, Krishnamurti L, Steinberg MH, Badesch DB, Gladwin MT; American Thoracic Society Ad Hoc Committee on Pulmonary Hypertension of Sickle Cell Disease. An official American Thoracic Society clinical practice guideline: diagnosis, risk stratification, and management of pulmonary hypertension of sickle cell disease. Am J Respir Crit Care Med. 2014 Mar 15;189(6):727-40. doi: 10.1164/rccm.201401-0065ST. PMID 24628312
- [Background] Barst RJ, Mubarak KK, Machado RF, Ataga KI, Benza RL, Castro O, Naeije R, Sood N, Swerdlow PS, Hildesheim M, Gladwin MT; ASSET study group*. Exercise capacity and haemodynamics in patients with sickle cell disease with pulmonary hypertension treated with bosentan: results of the ASSET studies. Br J Haematol. 2010 May;149(3):426-35. doi: 10.1111/j.1365-2141.2010.08097.x. Epub 2010 Feb 17. PMID 20175775
- [Background] Machado RF, Barst RJ, Yovetich NA, Hassell KL, Kato GJ, Gordeuk VR, Gibbs JS, Little JA, Schraufnagel DE, Krishnamurti L, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Onyekwere O, Castro OL, Sachdev V, Waclawiw MA, Woolson R, Goldsmith JC, Gladwin MT; walk-PHaSST Investigators and Patients. Hospitalization for pain in patients with sickle cell disease treated with sildenafil for elevated TRV and low exercise capacity. Blood. 2011 Jul 28;118(4):855-64. doi: 10.1182/blood-2010-09-306167. Epub 2011 Apr 28. PMID 21527519

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Macitentan
Started | 4
Completed | 1
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Macitentan
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: The occurrence of treatment emergent AEs includes having any of the following: vaso-occlusive crises requiring hospitalization; acute congestive heart failure; hypotension (defined as a mean arterial pressure less than 60mmHg); decrease in hemoglobin concentration by greater than 1 g/dL.
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Change in Right Arterial Pressure (RAP)
Description: RAP will be assessed by right heart catheterization. Normal range is 2-6 mmHg.
Time Frame: Baseline, 16 weeks
Measure: Number; unit: mmHg
Arm/Group | Macitentan
Number analyzed (Participants) | 1
mmHg | -5

3. Secondary Outcome: Change in Systolic Right Ventricular Pressure (RVSP)
Description: RVSP will be assessed by right heart catheterization. Normal range is 15-25 mmHg.
Time Frame: Baseline, 16 weeks
Measure: Number; unit: mmHg
Arm/Group | Macitentan
Number analyzed (Participants) | 1
mmHg | 3

4. Secondary Outcome: Change in Diastolic Pulmonary Artery Pressure (PADP)
Description: PADP will be assessed by right heart catheterization. Normal range is 8-15 mmHg.
Time Frame: Baseline, 16 weeks
Measure: Number; unit: mmHg
Arm/Group | Macitentan
Number analyzed (Participants) | 1
mmHg | -5

5. Secondary Outcome: Change in Systolic Pulmonary Artery Pressure (SPAP)
Description: SPAP will be assessed by right heart catheterization. Normal range is 15-25 mm Hg.
Time Frame: Baseline, 16 weeks
Measure: Number; unit: mmHg
Arm/Group | Macitentan
Number analyzed (Participants) | 1
mmHg | 7

6. Secondary Outcome: Change in Systemic Vascular Resistance Index (SVR)
Description: Systemic vascular resistance (SVR) will be assessed with this formula Systemic Vascular Resistance (SVR) = 80x(Mean Arterial Pressure - Mean Venous Pressure or CVP) / Cardiac Output. Normal range is 800 - 1200 dynes-sec/cm-5.
Time Frame: Baseline, Week 16
Measure: Number; unit: dynes-sec/cm-5.
Arm/Group | Macitentan
Number analyzed (Participants) | 1
dynes-sec/cm-5. | -528

7. Secondary Outcome: Change in Cardiac Index (CI)
Description: Cardiac index (CI) will be measured in L/min/m^2. The normal range for CI is 2.5 to 4 L/min/m^2.
Time Frame: Baseline to Week 16
Measure: Number; unit: L/min/m^2
Arm/Group | Macitentan
Number analyzed (Participants) | 1
L/min/m^2 | .23

8. Secondary Outcome: Change in 6 Minute Walk Distance (6MWD)
Description: The 6 minute walk test (6MWT) assesses distance walked over 6 minutes (6MWD) as a sub-maximal test of aerobic capacity/endurance. Participants will walk at their normal pace for 6 minutes.
Time Frame: Baseline, 16 weeks
Measure: Number; unit: meters
Arm/Group | Macitentan
Number analyzed (Participants) | 1
meters | -89

9. Secondary Outcome: Assess Change of Borg Dyspnea Index
Description: The Borg Dyspnea Index (BDI) is a 0 to 10 rated self reported numerical score used to measure dyspnea during submaximal exercise and will be administered immediately following the 6MWT. The higher the score, the more dyspnea.
Time Frame: Baseline, 16 weeks
Measure: Number; unit: score on a scale
Arm/Group | Macitentan
Number analyzed (Participants) | 1
score on a scale | 6

10. Secondary Outcome: World Health Organization (WHO) Functional Classification
Description: The WHO functional classification will be assessed and documented with the WHO Class.
  Class I Patients with pulmonary hypertension (PH) but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain or near syncope.
  Class II Patients with PH resulting in a slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III Patients with PH resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class IV Patients with PH with inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure. Dyspnea and/or fatigue may even be present at rest. Discomfort is increased by any physical activity.
  The Class is inversely related to function.
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Macitentan
Number analyzed (Participants) | 1
participants
  Class 1 | 0
  Class 2 | 0
  Class 3 | 1
  Class 4 | 0

11. Secondary Outcome: Change in NT-proB-type Natriuretic Peptide (NT-pro-BNP)
Description: The normal range for NT-pro-BNP is less than 300 picograms of BNP per milliliter (pg/ml) of blood; higher levels are less favorable.
Time Frame: Baseline, 16 weeks
Measure: Number; unit: pg/mL
Arm/Group | Macitentan
Number analyzed (Participants) | 1
pg/mL | 10528

12. Secondary Outcome: Change in Cardiac Output (CO)
Description: Cardiac output (CO) will be measured in L/min/m^2. The normal range for CO is 4 to 8 L/min/m^2.
Time Frame: Baseline, Week 16
Measure: Number; unit: L/min/m^2
Arm/Group | Macitentan
Number analyzed (Participants) | 1
L/min/m^2 | .29

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Macitentan
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=1)
nausea and vomiting (Gastrointestinal disorders) | 1 (6)

LIMITATIONS AND CAVEATS:
Early termination as unable to enroll participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT02651272/Prot_SAP_000.pdf